CLINICAL TRIAL: NCT04218123
Title: Assessing the Efficacy of a Serotonin and Norepinephrine Reuptake Inhibitor for Improving Meniere's Disease Outcomes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: American Hearing Research Foundation (Other); Cures Within Reach (Other)
Responsible Party: Principal Investigator, Habib Rizk,MD, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00091200
Record Dates: First submitted 2019-12-30; First posted 2020-01-06 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Meniere Disease
MeSH Terms: conditions — Meniere Disease | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Venlafaxine Arm (Experimental)
  Interventions: Drug: Venlafaxine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Venlafaxine — Daily oral intake 37.5 mg
  Arms: Venlafaxine Arm
Drug: Placebo oral tablet — Daily oral intake
  Arms: Placebo

SUMMARY:
As of yet, the cause of Meniere's disease is uncertain and there is no cure. Given the lack of high level evidence for treatments, we seek to perform a randomized, placebo-controlled, double-blind, crossover, pilot trial of venlafaxine for treating Meniere's disease. Venlafaxine is a safe and well-tolerated medication. It has never been trialed in Meniere's disease, but there is evidence that it could be effective in helping with vertigo attacks and other aspects of the disorder.

ELIGIBILITY:
Study subjects will be prospectively recruited from the population of patients presenting with dizziness to our tertiary, multidisciplinary, vestibular-focused, neurotology clinic. Subjects must meet the following inclusion criteria:

* be 18 years of age or older;
* have definite MD as defined by the Barany Society 2015 international consensus statement;
* have active MD with at least 2 vertigo episodes in the month prior to enrollment; and score at least 36 on the Dizziness Handicap Inventory (DHI), representing at least moderate handicap.

Patients with the following will be excluded:

* other concurrent vestibular or balance disorder (especially those with vestibular migraine-related vertigo episodes despite not meeting diagnostic criteria for vestibular migraine);
* currently taking venlafaxine, SSRIs, or SNRIs;
* history of medical (e.g. gentamicin) or surgical (e.g. labyrinthectomy) vestibular ablative treatment;
* history of otologic, lateral skull base, or brain surgery;
* history of radiation to the head or neck;
* known neurologic disorder affecting cognition;
* currently taking another serotonin modulating medication;
* seizures;
* stroke;
* myocardial infarction;
* hepatic or renal impairment;
* hyperlipidemia;
* coagulopathy;
* psychiatric disorder other than anxiety or depression;
* glaucoma;
* uncontrolled hypertension;
* pregnancy or intention of pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Habib Rizk, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical Univeristy of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rizk H, Monaghan NP, Shah S, Liu Y, Keith BA, Jeong S, Nguyen SA. Efficacy of a Serotonin-Norepinephrine Reuptake Inhibitor as a Treatment for Meniere Disease: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Nov 1;150(11):935-942. doi: 10.1001/jamaoto.2024.2241. PMID 39235772

RESULTS

PARTICIPANT FLOW:
Groups:
- Venlafaxine, Then Placebo: Venlafaxine 37.5mg tablet by mouth once daily in first 8 week period and placebo tablet by mouth once daily in the second 8 week period.
- Placebo, Then Venlafaxine: Placebo tablet by mouth once daily in first 8 week period and venlafaxine 37.5mg tablet by mouth once daily in the second 8 week period.
Period: Overall Study
Arm/Group | Venlafaxine, Then Placebo | Placebo, Then Venlafaxine
Started | 20 | 20
Completed | 18 | 20
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venlafaxine, Then Placebo | Placebo, Then Venlafaxine | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (17.2) | 58.3 (11) | 56.6 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Vertigo Episodes
Description: Patients will be keeping a diary throughout the study period and beyond.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of episodes
Groups:
- Venlafaxine Arm: Venlafaxine 37.5 mg tablet by mouth once daily
- Placebo Arm: Placebo tablet by mouth once daily
- Baseline Score: Baseline score upon enrollment in the study
Arm/Group | Venlafaxine Arm | Placebo Arm | Baseline Score
Number analyzed (Participants) | 40 | 40 | 40
number of episodes | 5.41 (4.44) | 5.03 (4.57) | 13.78 (10.05)
Statistical Analysis 1: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; Test type: Equivalence — p value <0.05 required to be considered nonequivalent; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Venlafaxine Arm vs Baseline Score; Test type: Equivalence — p value of <0.05 required for result to be considered nonequivalent; p < 0.05, ANOVA; Anova Post Hoc Analysis
Statistical Analysis 3: Comparison: Placebo Arm vs Baseline Score; Test type: Equivalence — p value of <0.05 required for result to be considered nonequivalent; p < 0.05, ANOVA; Anova Post Hoc Analysis
Statistical Analysis 4: Comparison: Venlafaxine Arm vs Placebo Arm; Test type: Equivalence — p value of <0.05 required for result to be considered nonequivalent; p > 0.05, ANOVA; Anova Post Hoc Analysis

2. Primary Outcome: Severity of Vertigo
Description: The study team will use a modified version of vertigo control classification because the treatment phases are 2 months long and the study team will not be able to wait 18-24 months after treatment to assess efficacy per academy guidelines. Previous studies have defined four categories of response to treatment: 1) very good response if more than 75% reduction in vertigo spells frequency and/or intensity, 2) good response if 50-75% reduction, 3) fair response if 25-50% reduction, and 4) poor response if less than 25% reduction.
  The vertigo classes will be defined as follows; Class A: 0 (complete control of vertigo) Class B: 0-40 or >60% reduction in mean vertigo episode severity (good control of vertigo) Class C: 41-80 or 20-60% reduction in severity (fair control of vertigo) Class D: 81-120 or -20-20% reduction in severity (no change in vertigo) Class E: >120 or >20% worsening in severity (worse vertigo)
Time Frame: 6 months
Measure: Number; unit: Percentage of members in arm
Arm/Group | Venlafaxine Arm | Placebo
Number analyzed (Participants) | 40 | 40
Percentage of members in arm
  Class A Control | 16 | 24
  Class B Control | 38 | 32
  Class C Control | 30 | 32
  Class D Control | 5 | 3
  Class E Control | 11 | 9

3. Secondary Outcome: Change in Score on The Medical Outcomes Study 20-item Short Form Health Survey
Description: The Medical Outcomes Study 20-item Short Form Health Survey is a 20-item general health questionnaire to assess quality of life in chronic diseases. It assesses 6 areas of health: physical functioning, role functioning, social functioning, mental health, health perceptions, and pain. Each score ranges between 0 and 100, with 100 indicating best possible function and 0 the worst possible function.
Time Frame: Baseline to end of treatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Arm | Placebo Arm | Baseline Score
Number analyzed (Participants) | 40 | 40 | 40
score on a scale
  Physical Functioning | 14.92 (3.34) | 14.54 (3.42) | 13.81 (3.6)
  Role Functioning | 4.62 (1.62) | 4.6 (1.61) | 4.38 (1.52)
  Mental Health | 22.24 (6.79) | 22 (5.95) | 20.95 (6.06)
  Social Functioning | 4.38 (1.67) | 4.54 (1.44) | 3.84 (1.44)
  Health Perceptions | 16.95 (4.91) | 16.17 (5.46) | 15.07 (5.1)
  Pain | 2.6 (1.44) | 2.74 (1.42) | 2.76 (1.52)
Statistical Analysis 1: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; SF20 Physical Functioning; Test type: Equivalence — p value <0.05 required to be considered nonequivalent; p = 0.31, ANOVA
Statistical Analysis 2: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; SF20 Role Functioning; Test type: Equivalence — p value of <0.05 required for result to be considered nonequivalent; p = 0.633, ANOVA
Statistical Analysis 3: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; SF20 Mental Health; Test type: Equivalence — p value of <0.05 required for result to be considered nonequivalent; p = 0.424, ANOVA
Statistical Analysis 4: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; SF20 Social Functioning; Test type: Equivalence — p value of <0.05 required for result to be considered nonequivalent; p = 0.057, ANOVA
Statistical Analysis 5: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; SF20 Health Perceptions; Test type: Equivalence — p value of <0.05 required for result to be considered nonequivalent; p = 0.296, ANOVA
Statistical Analysis 6: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; SF20 Pain; Test type: Equivalence — p value of <0.05 required for result to be considered nonequivalent; p = 0.872, ANOVA

4. Secondary Outcome: Change in Score on The Meniere's Disease Patient-Oriented Symptom Index (MDPOSI)
Description: The Meniere's Disease Patient-Oriented Symptom Index is a 23-item survey developed as a MD-specific tool to assess the impact of MD symptoms on patients' lives. The score ranges from 0 to 100 with the higher score indicating an active disease with significant impact on function and quality of life.
Time Frame: Baseline to end of treatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Arm | Placebo Arm | Baseline Score
Number analyzed (Participants) | 40 | 40 | 40
score on a scale | 46.81 (15.59) | 46.31 (16.32) | 50.68 (13.66)
Statistical Analysis 1: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; Test type: Equivalence — p value <0.05 required to be considered nonequivalent; p = 0.538, ANOVA

5. Secondary Outcome: Change in Score on Penn State Worry Questionnaire (PSWQ)
Description: The PSWQ is a 16-item survey for assessment of anxiety which has been used to identify generalized anxiety disorder. Scores range from 16 (Low worry) to 80 (high worry). A score higher than 60 is indicative of significant anxiety and risk for an anxiety disorder
Time Frame: Baseline to end of treatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Arm | Placebo Arm | Baseline Score
Number analyzed (Participants) | 40 | 40 | 40
score on a scale | 44.35 (14.36) | 45.63 (13.48) | 47.16 (14.11)
Statistical Analysis 1: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; Test type: Equivalence — p value <0.05 required to be considered nonequivalent; p = 0.686, ANOVA

6. Secondary Outcome: Change in Score on Patient Health Questionnaire (PHQ9)
Description: The Patient Health Questionnaire is a 9-item survey which assesses the severity of depression. A low score is indicative of little to no depressive symptoms, and a high score is indicative of Moderately severe to severe depressive symptoms. Scores range from 0 to 27 with scores higher than 20 indicative of significant risk for depression and scores below 10 indicative at most of a mild depression.
Time Frame: Baseline to end of treatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Arm | Placebo Arm | Baseline Score
Number analyzed (Participants) | 40 | 40 | 40
score on a scale | 5.49 (5.27) | 7.17 (5.73) | 7.43 (5.32)
Statistical Analysis 1: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; Test type: Equivalence — p value <0.05 required to be considered nonequivalent; p = 0.167, ANOVA

7. Secondary Outcome: Change in Score on Cognitive Failure Questionnaire (CFQ)
Description: The Cognitive Failure Questionnaire is a 25-item survey which assesses cognitive and executive function not tied to any specific disease state. It aims to assess perception, memory, and motor function in everyday tasks.The score ranges from 0 to 100 The higher score on the CFQ, the more frequent the cognitive failures experienced by the subject
Time Frame: Baseline to end of treatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Arm | Placebo Arm | Baseline Score
Number analyzed (Participants) | 40 | 40 | 40
score on a scale | 33.92 (16.35) | 36.4 (17.63) | 36.14 (18.18)
Statistical Analysis 1: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; Test type: Equivalence — p value <0.05 required to be considered nonequivalent; p = 0.8, ANOVA

8. Secondary Outcome: Change in Score on Neuropsychological Vertigo Inventory (NVI)
Description: The English version of the Neuropsychological Vertigo Inventory consists of 28-items with a 5-point Likert scale for each question. It is a cognitive assessment specific to patients with dizziness. The NVI assesses 7 domains of cognition: space perception, attention, time perception, memory, emotional, visual/ocular and motor. The score ranges from 0 to 140. The higher the score on the NVI the worse the cognitive function of the subject.
Time Frame: Baseline to end of treatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Venlafaxine Arm: Venlafaxine 37.5mg tablet by mouth once daily
Arm/Group | Venlafaxine Arm | Placebo Arm | Baseline Score
Number analyzed (Participants) | 40 | 40 | 40
score on a scale | 59.41 (18.67) | 63.31 (17.78) | 65.11 (20.01)
Statistical Analysis 1: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; Test type: Equivalence — p value <0.05 required to be considered nonequivalent; p = 0.425, ANOVA

9. Secondary Outcome: Change in Score on Dizziness Handicap Inventory (DHI)
Description: The Dizziness Handicap Inventory is a 25-item questionnaire of self-perceived handicap from dizziness.There are 7 questions in the physical domain, 9 in the emotional domain, and 8 in the functional domain. It is scored from 0 (no perceived disability) to 100 (maximum perceived disability).
Time Frame: Baseline to end of treatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Arm | Placebo Arm | Baseline Score
Number analyzed (Participants) | 40 | 40 | 40
score on a scale | 45.46 (24.2) | 45.2 (20.77) | 55.62 (16.73)
Statistical Analysis 1: Comparison: Venlafaxine Arm vs Placebo Arm vs Baseline Score; Test type: Equivalence — p value <0.05 required to be considered nonequivalent; p = 0.054, ANOVA

ADVERSE EVENTS:
Time Frame: 22 weeks
Arm/Group | Venlafaxine Arm | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 6/40 | 3/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Venlafaxine Arm (N=40) | Placebo (N=40)
Dry mouth (General disorders) | 1 | 1
Nausea/vomiting (Gastrointestinal disorders) | 4 | 0
Decreased Appetite (General disorders) | 1 | 1
Insomnia (General disorders) | 0 | 1
Decreased Energy (General disorders) | 0 | 1
Sweating (General disorders) | 1 | 1
Weight Change (General disorders) | 0 | 1
Tinnitus (Nervous system disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was designed in 2019 with a power analysis that estimated a 20% placebo response in Meniere's Disease. This was a gross underestimation in hindsight. A systematic review with meta-analysis published in 2023 has illustrated that this effect is much stronger, closer to 50% in patients with Meniere's Disease, which may affect the ability to detect symptomatic differences between venlafaxine and placebo treatment periods, respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT04218123/Prot_SAP_001.pdf